CLINICAL TRIAL: NCT07096609
Title: A Single-center, Single-arm Phase II Study to Evaluate the Efficacy and Safety of Lenvatinib in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) Who Have Failed Treatment With Imatinib, Sunitinib, and Regorafenib
Brief Title: Lenvatinib After Progression on Imatinib, Sunitinib, and Regorafenib for GIST Patients
Acronym: LONGIST
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jaewon Hyung, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2502
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: GIST
Keywords: GIST; Lenvatinib
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib treatment (Experimental)
  Interventions: Drug: Lenvatinib Capsules

INTERVENTIONS:
Drug: Lenvatinib Capsules — Lenvatinib will be administered orally once daily at a dose of 12 mg (for patients weighing ≥ 60 kg) or 8 mg (for patients weighing < 60 kg). Each treatment cycle consists of 4 weeks (i.e., 28 days).

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of lenvatinib in patients with metastatic or advanced GIST who have failed at least imatinib, sunitinib, and regorafenib treatment.

DETAILED DESCRIPTION:
The discovery of KIT gene mutations and the development of the KIT tyrosine kinase inhibitor imatinib (Glivec™, Novartis) have significantly improved the survival rates of patients with advanced and metastatic gastrointestinal stromal tumors (GIST). More recently, sunitinib (Sutene™, Pfizer) and regorafenib (Stivarga®, Bayer) have been proven effective as second- and third-line therapies, respectively, for patients who have failed imatinib treatment. However, nearly all patients eventually develop resistance to first-line imatinib, second-line sunitinib, and third-line regorafenib, resulting in disease progression. Although ripretinib, a fourth-line treatment, has demonstrated an improvement in progression-free survival to 6.3 months compared to placebo in the phase III INVICTUS trial, it remains inaccessible in many regions, including Korea, limiting its clinical application. Therefore, there is an urgent need for new therapeutic alternatives after imatinib, sunitinib, and regorafenib in clinical practice.

Lenvatinib is a multi-targeted tyrosine kinase inhibitor with potent anti-angiogenic activity, primarily targeting VEGFR1-3 with IC₅₀ values of 4.7, 3.0, and 2.3 nmol/L, respectively. It also exhibits inhibitory activity against c-KIT (IC₅₀: 85 nmol/L) and PDGFR-α (IC₅₀: 29 nmol/L). Pharmacokinetically, lenvatinib is rapidly absorbed with a bioavailability of 85% and has an elimination half-life of approximately 28 hours. The LENVAGIST study, presented at ESMO 2024, was a phase II randomized, placebo-controlled trial that demonstrated the significant clinical activity of lenvatinib in patients with advanced GIST who had progressed after treatment with imatinib and sunitinib. In this study, the 4-month progression-free survival rate was 39% in the lenvatinib group versus 11% in the placebo group (HR 0.44; 95% CI 0.27-0.71; p=0.0008), and the median overall survival was 14.4 months versus 8.7 months, respectively. Treatment-related grade ≥3 adverse events were observed in 56.4% of patients in the lenvatinib group and 18.4% in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years at the time of providing written informed consent.
2. Histologically confirmed metastatic and/or advanced (unresectable or recurrent) GIST with positivity for CD117(+), DOG-1(+), or harboring mutations in the KIT or PDGFRα genes.
3. Documented failure of prior treatment with imatinib, sunitinib, and regorafenib due to disease progression and/or intolerance.

   * Note: There is no limitation on the number of prior therapies. Prior use of other tyrosine kinase inhibitors (TKIs) or chemotherapy in combination with imatinib, sunitinib, or regorafenib is permitted.
   * Disease progression is defined as:

     1. Increase in tumor size by ≥ 20% per mRECIST version 1.1
     2. Emergence of unequivocal new lesions (excluding newly developed small cystic liver lesions within 6 months after initiation of TKI treatment)
     3. Appearance of new solid nodules within cystic masses
     4. Increase in the size of existing solid nodules within cystic masses (>20%)
   * Intolerance to prior TKIs is defined as:

     1. Drug compliance <75% due to ≥ Grade 2 non-hematologic toxicity, despite dose reduction to one level below the standard dose (i.e., imatinib 300 mg/day; sunitinib 37.5 mg/day on a 4-week on/2-week off schedule or 25 mg/day on a continuous schedule; regorafenib 120 mg/day)
     2. Despite the same dose reduction as above, the occurrence of febrile neutropenia, Grade 4 neutropenia lasting more than 6 days, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with clinically significant bleeding, or Grade 3-4 or persistent ≥ Grade 2 non-hematologic toxicity deemed intolerable
4. ECOG performance status of 0-2.
5. All toxicities from previous treatments must have recovered to Grade 0 or 1 as per NCI-CTCAE version 5.0.
6. At least one measurable lesion as defined by mRECIST version 1.1.
7. Adequate bone marrow, liver, renal, and other organ function:

   * Absolute neutrophil count (ANC) ≥ 1,500/mm³
   * Platelets ≥ 100,000/mm³
   * Hemoglobin ≥ 8.0 g/dL
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * AST/ALT ≤ 2.5 × ULN (or ≤ 5 × ULN in case of liver metastases)
   * Serum creatinine ≤ 1.5 × ULN
8. Life expectancy ≥ 12 weeks
9. A washout period equivalent to at least 4 times the half-life of previous TKI or chemotherapeutic agents is required(Imatinib and regorafenib: ≥ 1 week; Sunitinib: ≥ 2 weeks)
10. Signed written informed consent

Exclusion Criteria:

1. Women of childbearing potential who are pregnant or breastfeeding
2. Women or men unwilling to use effective contraception during the study treatment period and for 6 months after the last dose of the investigational drug
3. All participants (both men and women) must use barrier contraception during the treatment period and for at least 1 month after the final dose
4. Women of childbearing potential are defined as sexually mature females who have not undergone hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., had menstruation within the past 12 months)
5. History of any of the following within 6 months prior to enrollment: myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass surgery, congestive heart failure classified as NYHA Class III or IV, stroke or transient ischemic attack (TIA), or clinically significant arrhythmias requiring treatment
6. Uncontrolled active infection
7. Diabetes mellitus with clinically significant signs of peripheral vascular disease
8. Acute or chronic liver disease, or any chronic hepatic disorder (patients with stable chronic hepatitis B are eligible)
9. Uncontrolled gastrointestinal toxicities greater than Grade 2 according to NCI-CTCAE (e.g., nausea, diarrhea, vomiting)
10. Any severe acute or chronic medical or psychiatric condition, or clinically significant abnormal laboratory finding, that may increase the risk associated with study participation or investigational drug administration, or interfere with the interpretation of study results, as determined by the investigator
11. History of life-threatening bleeding or any Grade 3 or 4 bleeding event requiring transfusion, endoscopic intervention, or surgical procedure within 3 months prior to initiation of study drug
12. Treatment with clinically significant systemic anticoagulant or antithrombotic agents within 7 days prior to consent that, in the opinion of the investigator, may put the patient at risk. Use of aspirin is permitted up to a maximum dose of 325 mg/day
13. Uncontrolled hypertension (blood pressure ≥ 140/90 mmHg) that is not adequately managed with medication, or change in antihypertensive regimen within 7 days prior to consent; such patients may be at increased risk during VEGF inhibitor therapy
14. Major surgery, significant trauma (e.g., bone fracture), or non-healed wounds within 3 weeks prior to consent (procedures such as catheter insertion are not considered major)
15. History of other significant cardiovascular or vascular conditions within 6 months prior to consent that, in the opinion of the investigator, may place the patient at risk during VEGF inhibitor therapy, including but not limited to hypertensive crisis, hypertensive encephalopathy, stroke, transient ischemic attack (TIA), or clinically significant peripheral vascular disease
16. Clinically significant glomerulonephritis, biopsy-proven tubulointerstitial nephritis, crystal nephropathy, or other history of renal failure
17. Known diagnosis of HIV infection (HIV testing is not mandatory)
18. History of another primary malignancy that has recently become clinically significant or currently requires active intervention
19. Evidence of brain metastasis on radiological imaging (e.g., CT or MRI) in patients presenting with symptoms suggestive of central nervous system involvement
20. History of alcohol or substance abuse disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DCR(disease control rate) at 12 weeks | at 12 weeks
  To evaluate the disease control rate (DCR; defined as the sum of partial responses and stable disease) at 12 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No